CLINICAL TRIAL: NCT04517565
Title: Longitudinal Neuroimaging in Sturge-Weber Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Csaba Juhasz, Professor, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sturge-Weber neuroimaging
Record Dates: First submitted 2020-08-07; First posted 2020-08-18 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Sturge-Weber Syndrome
MeSH Terms: conditions — Sturge-Weber Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with SWS or high-risk facial port-wine birthmark (Experimental): All patients with SWS brain involvement (based on previous imaging) or facial port-wine birthmark indicating a high risk for SWS brain involvement will undergo a brain MRI and neuro-psychology testing.
  Interventions: Diagnostic Test: Brain magnetic resonance imaging; Behavioral: Neuro-psychology testing

INTERVENTIONS:
Diagnostic Test: Brain magnetic resonance imaging — Brain magnetic resonance imaging (MRI) will be done using multiple sequences to evaluate presence, type and severity of brain abnormalities in enrolled subjects.
  Other Names: MRI
Behavioral: Neuro-psychology testing — Participants will undergo age-appropriate neuro-psychology testing to assess motor, language and other neuro-cognitive functions potentially affected by Sturge-Weber syndrome.
  Other Names: neuro-cognitive testing; neuro-psychology

SUMMARY:
In this project the accuracy of a novel, rapid magnetic resonance imaging (MRI) approach to detect brain abnormalities in patients with Sturge-Weber syndrome (SWS) will be tested; this new imaging approach, that can create multiple types of MR images in about 5 minutes, without contrast administration (and sedation even in young children), can be also readily applied in other pediatric brain disorders in the future. The investigators will also study how advanced MRI, including susceptibility-weighted and diffusion tensor imaging can detect detailed signs of brain vascular and neuronal reorganization that helps improve neurological and cognitive outcome of children and young adults with SWS, who could benefit from targeted interventions in the future to minimize neurocognitive deficits in affected patients. All enrolled subjects will undergo advanced brain MRI and neurocognitive evaluation to achieve these goals.

DETAILED DESCRIPTION:
This project will combine advanced neuroimaging with detailed neuro-psychology evaluation, performed in both children and young adults affected by Sturge-Weber syndrome, in order to address two main aims, each of them with two research hypotheses:

AIM 1. To determine the accuracy of a novel, rapid MRI approach for detection of early and advanced SWS brain abnormalities as compared to a standard MRI acquisition (current clinical standard).

Hypothesis 1.1. In young children with SWS, rapid MRI using STAGE will detect the presence and extent of brain involvement with high accuracy when compared to standard MRI.

Hypothesis 1.2. In children, adolescents, and young adults, rapid MRI using STAGE will have high accuracy to detect advanced brain vascular and parenchymal abnormalities as compared to standard MRI.

Since the detrimental neurocognitive effects of SWS brain involvement are most robust during the early disease course, early interventions, including preventive antiepileptic treatment in children with high-risk port-wine birthmark are being considered. This paradigm changing therapeutic approach would greatly benefit from safe, accurate imaging for rapid screening not requiring sedation or contrast injection. In this aim, the investigators will evaluate a recently developed, rapid, multi-echo MRI acquisition protocol (STAGE: Strategically Acquired Gradient Echo) for its ability to detect early and late SWS-related vascular and brain tissue abnormalities.

AIM 2. To assess the role of key vascular and neuronal compensatory mechanisms in neurocognitive outcome in unilateral SWS.

Hypothesis 2.1. Extensive ipsilateral deep vein collaterals will protect the SWS-affected hemisphere as indicated by relatively preserved structural brain integrity and global neurocognitive functions.

Hypothesis 2.2. In unilateral SWS, reorganized structural networks in the contralateral cerebral hemisphere will predict alterations in specific cognitive, motor, language, and executive functions.

Recent studies revealed two, potentially powerful compensatory mechanisms that may offset the effects of SWS-related brain injury in unilateral SWS: (i) expanding ipsilateral deep venous collaterals, and (ii) contralateral brain reorganization associated with preserved verbal functions at the cost of non-verbal abilities ("crowding" effect) in left-hemispheric SWS. Here the investigators will use advanced MRI techniques (such as susceptibility-weighted and diffusion tensor imaging (DTI)-based connectome analysis) to evaluate the long-term global and specific neurocognitive effects of venous vascular remodeling and structural reorganization, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with Sturge-Weber syndrome (SWS):

   1. Age 3 months - 30 years;
   2. Presence of a facial port-wine birthmark (PWB) indicating a risk for SWS and/or evidence of SWS brain involvement based on the presence of one or more intracranial SWS brain abnormalities from previous clinical imaging (MRI or computed tomography) scan(s) with or without a facial PWB. SWS brain abnormalities can include both brain vascular and/or parenchymal abnormalities (including atrophy, calcification, etc.);
   3. In children who will undergo formal neuropsychology testing including detailed language testing (age 3 years and above): proficiency of English language.
2. Healthy control subjects:

   1. Age 3 years - 30 years;
   2. No history of neurological or psychiatric disorder

Exclusion Criteria:

For all subjects:

1. Metal in the head or mouth that would preclude safe, artifact-free MRI scanning; or any other metal or electronic device contraindicated for MRI scanning.
2. History of severe claustrophobia, precluding staying still in the scanner for up to 30 minutes.
3. Pregnancy (pregnant women will be scheduled for the study after delivery).

For SWS subjects, who will receive MRI contrast material, additional exclusion criteria:

1. History of sensitivity to MRI contrast material;
2. History of renal disease that would preclude safe administration of MRI contrast material

Ages: 3 Months to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Accuracy of detection of Sturge-Weber syndrome brain involvement by a novel fast magnetic resonance imaging (MRI) approach as compared to standard MRI. | During procedure
  Presence (score 1) vs. absence (score 0) of SWS brain abnormalities in each of 8 cerebral lobes using fast MRI compared with the same scores obtained from standard MRI, obtained in the same imaging session, as the ground truth.
Correlation of enlarged cerebral deep vein scores, measured by magnetic resonance imaging (MRI), with full scale IQ acquired within 1 day. | 1 day
  Full scale IQ (normal mean: 100, standard deviation: 15) will be determined and its correlation with enlarged deep vein scores (range: 0-12, 0 indicating no enlarged deep veins, 12 indicating the most extensive enlarged deep veins) measured by MRI calculated.
Correlation of diffusion tensor imaging (DTI) brain connectivity score with verbal IQ acquired within 1 day. | 1 day
  Verbal IQ (normal mean: 100, standard deviation: 15) will be determined by neuropsychology evaluation and correlated with DTI brain connectivity scores (range: 0-1, 0 indicating no connectivity, 1 indicating the strongest connectivity) measured by MRI.
Correlation of diffusion tensor imaging (DTI) brain connectivity score with non-verbal IQ acquired within 1 day. | 1 day
  Non-verbal IQ (normal mean: 100, standard deviation: 15) will be determined by neuropsychology evaluation and correlated with DTI brain connectivity scores (range: 0-1, 0 indicating no connectivity, 1 indicating the strongest connectivity) measured by MRI.

SECONDARY OUTCOMES:
Correlation of enlarged deep vein scores determined by magnetic resonance imaging (MRI) with motor scores acquired within 1 day. | 1 day
  Motor scores (normal mean: 100, standard deviation: 15), determined during neuro-psychology evaluation, will be correlated with enlarged deep vein scores (range: 0-12, 0 indicating no enlarged deep veins, 12 indicating the most extensive enlarged deep veins) determined by MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University / Children's Hospital of Michigan, Detroit, Michigan, United States